CLINICAL TRIAL: NCT01213927
Title: CIRRAL: Hepatocellular Carcinoma in Patients With Uncomplicated Alcoholic Cirrhosis: Incidence and Predictive Factors. A Multicentric Prospective Cohort
Brief Title: National Cohort of Uncomplicated Alcoholic Cirrhosis
Acronym: CIRRAL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI09020
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Alcoholic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At enrollement, 20 ml of blood will be collected for freezing and storage of serum and plasma, and constitution of a DNA library
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hepatocellular carcinoma (HCC) is a major public health problem, whose incidence is increasing in developed countries and is the leading cause of death in patients with cirrhosis. The diagnosis and the early management are key issues that could improve the prognosis. In France, alcoholic cirrhosis is the leading cause of HCC, while the aetiology of underlying chronic liver disease is mainly hepatitis C (HCV) in Southern Europe and Japan, and hepatitis B (HBV) in Asia and Africa. In the next years, due to the improved results of anti-viral therapies, this trend should be reinforced with a decreasing proportion of HCC related to viral cirrhosis and an increasing proportion of HCC related to alcoholic cirrhosis. However, natural history of alcoholic cirrhosis remains poorly understood, most studies being retrospective and including a small number of patients. This project is filed by the consortium CIRRAL including French Academic hospitals centers currently involved and referees in the field of alcoholic liver disease and HCC (8 at the moment, and more in the next months). It is a national multicenter prospective study that will include 1200 patients with alcoholic cirrhosis histologically proven over 3 years. The main goal of this cohort is to describe the natural history of a large number of patients with alcoholic cirrhosis prospectively followed, and to identify predictors of the occurrence of HCC.

DETAILED DESCRIPTION:
Patients will be selected for the study if they met all the inclusion criteria, without any of the non-inclusion criteria, ie compensated Child Pugh A alcoholic cirrhosis without viral chronic hepatitis B or C, and without any detectable HCC. They will be offered, during a consultation as part of their usual care, to participate in the study. An information note will be issued. Patients agreeing to participate should date and sign informed consent. Usual biological tests and liver ultrasonography will be performed if not done within 90 days prior to inclusion. During this visit, 20 ml of blood will be collected for freezing and storage of serum and plasma, and constitution of a DNA library.

From the reviews conducted at baseline, patients with at least one exclusion criteria (ie decompensation of cirrhosis, Child Pugh score ≥ 7, co-infection with HBV or HCV, or liver focal lesion suggestive of HCC will be excluded (and their serum samples achieved for the BioBank will be destroyed):

Monitoring: According to current guidelines, patients will have periodical surveillance with liver ultrasonography and medical consultation at least every 6 months, blood tests at least every year, periodic assessment of esophageal and gastric varices (every 1 to 3 years) and prevention of their rupture if any. An additional blood sampling of 20 ml will be taken at baseline and every year in order to perform serum, plasma, and DNA libraries; Data will be standardized and centralized in a single database.

Statistical Analysis: Methods for censored data with competitive risks. Number of subjects to include: The planned number is 1200 subjects included in 3 years. Assuming a minimal annual incidence of HCC about 2% in patients with alcoholic cirrhosis, and a proportion of lost to follow-up of around 20% in this poorly compliant population, a sample of 3000 patients could demonstrate the existence of predictive factors for the occurrence of HCC associated with a relative risk at least equal to 2, with a power of 90%. However, the enrollment of 3000 patients recruited in three years is not a realistic goal. For practical reasons and since the data currently available are very limited regarding the precise incidence of HCC and the strength of association between risk factors and HCC in patients with alcoholic cirrhosis, the minimum number of patients included in the cohort CIRRAL was set at 1200. Regarding an expected percentage of patients lost to follow close to 20%, the final number of patients with sufficient follow-up will be 1000.

Expected results

1. description of the incidence of HCC occurrence in patients with alcoholic cirrhosis;
2. identification of predictive factors for the occurrence of HCC c) identification of prognostic factors for survival. In addition, nested scientific projects will use the database and collected samples of this prospective cohort, thus constituting significant savings of resources. However, these nested scientific projects should include a specific need of organization and financing clean, and may involve only a fraction of the population included. The areas involved are very varied (immunology, genetics, imaging, evaluation of fibrosis, biostatistics, , quality of life, economy, etc.).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* histologically proven cirrhosis
* no previous HCC (treated or not )
* excessive consumption of alcohol, considered as the main cause of cirrhosis
* signed informed consent.

Exclusion Criteria:

* serious associated short-term life threatening disease (except associated HIV viral infection and the liver disease itself),
* decompensation of cirrhosis (bleeding or ascites),
* co-infection with HBV or HCV;
* liver focal lesion suggestive of HCC
* Child Pugh score ≥ 7 (Class B or C).
* patient under guardianship
* pregnant women
* inability to regular monitoring, for whatever reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French primary care hospitals
Sampling Method: Non-Probability Sample
Enrollment: 709 (Actual)
Dates: Start 2010-10; Primary Completion 2018-11 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
HCC Occurrence | 3 years
  cumulative incidence within 3 years

SECONDARY OUTCOMES:
Mortality | 3 years
  overall mortality - whatever the cause of death
Liver-related mortality | 3 years
  cumulative incidence of liver-related deaths
Alcohol- and cirrhosis-related event free survival | 3 years
  event free survival where events are ascitis, digestive hemorrhage, icterus, encephalopathy, non-liver events related to alcohol, bacterial infection and death free of those events

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie GANNE, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Jean Verdier hospital (AP-HP), Bondy, France

REFERENCES:
- [Derived] Louvet A, Bourcier V, Archambeaud I, d'Alteroche L, Chaffaut C, Oberti F, Moreno C, Roulot D, Dao T, Moirand R, Duclos-Vallee JC, Goria O, Nguyen-Khac E, Pol S, Carbonell N, Gournay J, Elkrief L, Fouchard-Hubert I, Chevret S, Ganne-Carrie N; CIRRAL group. Low alcohol consumption influences outcomes in individuals with alcohol-related compensated cirrhosis in a French multicenter cohort. J Hepatol. 2023 Mar;78(3):501-512. doi: 10.1016/j.jhep.2022.11.013. Epub 2022 Nov 22. PMID 36423805
- [Derived] Ganne-Carrie N, Nahon P, Chaffaut C, N'Kontchou G, Layese R, Audureau E, Chevret S; CIRRAL group; ANRS CO12 CirVir group. Impact of cirrhosis aetiology on incidence and prognosis of hepatocellular carcinoma diagnosed during surveillance. JHEP Rep. 2021 Mar 26;3(3):100285. doi: 10.1016/j.jhepr.2021.100285. eCollection 2021 Jun. PMID 34522876